CLINICAL TRIAL: NCT04256369
Title: Rate of Termination of Commercial Premixed Parenteral Nutrition (PN) in Surgical Patients Secondary to High Serum Electrolyte Levels
Brief Title: Rate of Termination of Premixed Parenteral Nutrition (PN) in Surgical Patients Secondary to High Serum Electrolytes
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Hakeam Abdulaziz Hakeam, Clinical Pharmacy Specialist, Surgery. Pharmaceutical Care Division, King Faisal Specialist Hospital & Research Centre. Adjunct Assistant Clinical Professor College of Medicine, Alfaisal University., King Faisal Specialist Hospital & Research Center
Other Study IDs: 2191316
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Hyperphosphatemia; Hyperkalemia; Hypermagnesemia; Hypercalcemia
Keywords: Parenteral Nutrition; Hyperkalemia; Hypermagnesemia; Hyperphosphatemia; Hypercalcemia
MeSH Terms: conditions — Hyperphosphatemia; Hyperkalemia; Hypercalcemia; Hyperphagia | interventions — Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary Cohort: Starting premixed Olimel N9E and follow for electrolyte irregularities.
  Interventions: Combination Product: Parenteral Nutrition (PN) Premixed Olimel N9E

INTERVENTIONS:
Combination Product: Parenteral Nutrition (PN) Premixed Olimel N9E — Parenteral nutrition
  Other Names: Olimel N9E

SUMMARY:
Introduction:

Various commercial premixed parenteral nutrition (PN) solutions have been introduced to clinical practice in 3-compartment large volume bags. Olimel N9E is the formulary premixed PN formula at King Faisal Specialist Hospital and Research Centre (KFSH & RC). The commercial premixed PN was associated with a significant cost reduction compared to the compounded PN, with lower incidence of infectious complications, compared to the compounded PN formula. Electrolyte irregularities are commonly encountered with PN use. Patients who develop high serum potassium, magnesium or phosphate levels while receiving premixed PN are shifted to a compounded PN with lower electrolyte content. This study aims to describe the incidence of shifting of premixed PN to a compounded PN secondary to high serum electrolytes in surgical patients receiving commercial premixed PN.

Methods:

This is a prospective, cohort, study, to be conducted at KFSH & RC, Riyadh. This study is proposed to commence after obtaining the approval of the Research Ethical Committee at KFSH & RC. Patients enrolment will start after the approval at KFSH & RC, by data collection phase, that might extend for a suspected 6-month until achieving the target sample size of 55 patients. The analysis phase will follow and elapse for 2 months. This is followed by 2 months to get the initial abstract. All patients will have their potassium, magnesium, calcium and phosphorus levels assessed daily in the morning for the first 7 days of PN initiation. After the first week of PN support, according to the routine laboratories, electrolytes will be assessed at a minimum of three times a week thereafter while on PN. There will be no extra laboratory work obtained for the study purpose. The incidence of shifting from premixed PN to compounded PN will be assessed and reported. A description of the characteristics of patients who develop high serum level of electrolytes will be undertaken using regression analysis.

DETAILED DESCRIPTION:
Methods Study design and centres This is a prospective, cohort, multi-centre study, to be conducted at King Faisal Specialist Hospital and Research Centre, (KFSH & RC), Riyadh. The study has been approved by KFSH&RC Office of Research Affairs representing the institutional review board (IRB).

Subjects:

Sample Size Sample size has been calculated using Raosoft website based on the total surgical patients who receive PN support on monthly bases, which is 20 patients per month, and the duration of the data collection is expected to elapse 6 months. This makes the field population represented by 120 patients. According to a previous study that assessed need for bolus of electrolytes, 7% of the eligible patients are expected to have the outcome. Allowing for 5% margin of error and 95% confidence level the target sample size will be 72 patients from KFSH&RC. Collaborating centers withdrew from this study due to insufficient eligible patients given the COVID-19 pandemic.

Protocol Surgical patients starting PN will be screened for the inclusion and exclusion criteria by the investigators of the study. Eligible patients will be asked to sign a consent form.

All patients will start PN after normalization of the following electrolytes potassium, magnesium, and phosphorus according to standard. Premixed PN formula, Olimel N9E will be started at a rate of 45 mL per hour for all patients on day 1 of PN support. After the routine assessment by pharmacists, the PN rate will be increased at an increment of 10 mL per hour on daily basis, representing the target goal of protein of 2 gm per kg according to the ideal body weight (IBW) , is achieved. Patients enrolled in the study will be followed while on PN support until cessation of PN or after 30 days of support have elapsed.

All patients will get their potassium, magnesium, and phosphorus levels assessed daily in the morning for the first 7 days of PN initiation. After the first week of PN support, electrolytes will be assessed at a minimum of three times a week thereafter while on PN. High electrolyte levels that develop on the following day of their respective low levels and corrected with bolus will not be considered as induced by PN.

Patients who develop hyperphosphatemia, hypermagnesemia, hyperkalaemia will get their PN stopped immediately and replaced with dextrose 10% water solution to run at 50 mL per hour till 21:00.Premixed PN will commence again at the same rate of the corresponding day. Patients who develop a second episode of any hyperphosphatemia, hypermagnesemia, or hyperkalaemia on the preceding day obtained from a blood sample will be shifted to the compounded PN.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted under the care of non-cardiac surgical services, whether planned for surgery or to manage a surgical complications that developed within 30 after surgery.
* Patients under the care of the following surgical teams: colorectal surgery, oncology surgery, general surgery, and thoracic surgery.
* Patients starting PN as a sole source for nutrition with feeding status is nil per os (NPO)
* Patients who receive sips of water or oral tablets will be included in this study.

Exclusion Criteria:

* Any degree of renal impairment defined as glomerular filtration rate < 60 mL/min/m2 as calculated according to the modification of diet in renal disease (MDRD) equation
* Morbid obesity defined as body mass index (BMI) of > 40 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥ 18) patients admitted to King Faisal Specialist Hospital and Research Centre, Riyadh , under non-cardiac surgical services, whether planned for surgery or to manage a surgical complication that developed within 30 after surgery, in which parenteral nutrition is indicated and is the sole source of nutrition.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of shifting of Olimel N9E premixed formula to compounded PN secondary to the development of elevated electrolyte levels in surgical patients receiving PN. | Until cessation of parenteral nutritional support or after 30 days of PN support have elapsed.
  Serum phosphate level of > 1.45 mmol/L, serum potassium level > 5.0 mmol/L, and serum magnesium level > 1.0 mmol/L.

SECONDARY OUTCOMES:
Rate of high serum levels of phosphate, magnesium, calcium, and potassium. | Until cessation of parenteral nutritional support or after 30 days of PN support have elapsed
  serum phosphate level of > 1.45 mmol/L, serum potassium level > 5.0 mmol/L, and serum magnesium level > 1.0 mmol/L
Risk factors associated with the development of hyperphosphatemia | Until cessation of parenteral nutritional support or after 30 days of PN support have elapsed
  Serum phosphate level of > 1.45 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Hakeam Hakeam, MS Pharm, Principal Investigator — King Faisal Specialist Hospital and Research Centre (KFSH&RC)
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
On publication, according to the journal requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After November 2020.
Access Criteria: Pending

REFERENCES:
- [Background] Maisonneuve N, Raguso CA, Paoloni-Giacobino A, Muhlebach S, Corriol O, Saubion JL, Hecq JD, Bailly A, Berger M, Pichard C. Parenteral nutrition practices in hospital pharmacies in Switzerland, France, and Belgium. Nutrition. 2004 Jun;20(6):528-35. doi: 10.1016/j.nut.2004.03.020. PMID 15165615
- [Background] Hall JW. Safety, cost, and clinical considerations for the use of premixed parenteral nutrition. Nutr Clin Pract. 2015 Jun;30(3):325-30. doi: 10.1177/0884533615578459. Epub 2015 Apr 10. PMID 25862011
- [Background] DeLegge MH. Parenteral nutrition therapy over the next 5-10 years: where are we heading? JPEN J Parenter Enteral Nutr. 2012 Mar;36(2 Suppl):56S-61S. doi: 10.1177/0148607111435333. Epub 2012 Feb 2. PMID 22301323
- [Background] Pontes-Arruda A, Zaloga G, Wischmeyer P, Turpin R, Liu FX, Mercaldi C. Is there a difference in bloodstream infections in critically ill patients associated with ready-to-use versus compounded parenteral nutrition? Clin Nutr. 2012 Oct;31(5):728-34. doi: 10.1016/j.clnu.2012.03.004. Epub 2012 May 8. PMID 22572624
- [Background] Berlana D, Almendral MA, Abad MR, Fernandez A, Torralba A, Cervera-Peris M, Pineiro G, Romero-Jimenez R, Vazquez A, Ramirez E, Yebenes M, Munoz A. Cost, Time, and Error Assessment During Preparation of Parenteral Nutrition: Multichamber Bags Versus Hospital-Compounded Bags. JPEN J Parenter Enteral Nutr. 2019 May;43(4):557-565. doi: 10.1002/jpen.1436. Epub 2018 Aug 29. PMID 30156305
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Background] Hardy G, Puzovic M. Formulation, stability, and administration of parenteral nutrition with new lipid emulsions. Nutr Clin Pract. 2009 Oct-Nov;24(5):616-25. doi: 10.1177/0884533609342445. PMID 19841249
- [Background] Biesalski HK, Bischoff SC, Boehles HJ, Muehlhoefer A; Working group for developing the guidelines for parenteral nutrition of The German Association for Nutritional Medicine. Water, electrolytes, vitamins and trace elements - Guidelines on Parenteral Nutrition, Chapter 7. Ger Med Sci. 2009 Nov 18;7:Doc21. doi: 10.3205/000080. PMID 20049067
- [Background] Boullata JI, Gilbert K, Sacks G, Labossiere RJ, Crill C, Goday P, Kumpf VJ, Mattox TW, Plogsted S, Holcombe B; American Society for Parenteral and Enteral Nutrition. A.S.P.E.N. clinical guidelines: parenteral nutrition ordering, order review, compounding, labeling, and dispensing. JPEN J Parenter Enteral Nutr. 2014 Mar-Apr;38(3):334-77. doi: 10.1177/0148607114521833. Epub 2014 Feb 14. PMID 24531708
- [Background] Beattie C, Allard J, Raman M. Comparison Between Premixed and Compounded Parenteral Nutrition Solutions in Hospitalized Patients Requiring Parenteral Nutrition. Nutr Clin Pract. 2016 Apr;31(2):229-34. doi: 10.1177/0884533615621046. Epub 2016 Feb 17. PMID 26888855
- [Background] Fantoni D, Shih AC. Perioperative Fluid Therapy. Vet Clin North Am Small Anim Pract. 2017 Mar;47(2):423-434. doi: 10.1016/j.cvsm.2016.11.004. PMID 28164837
- [Background] Peppers MP, Geheb M, Desai T. Endocrine crises. Hypophosphatemia and hyperphosphatemia. Crit Care Clin. 1991 Jan;7(1):201-14. PMID 2007215
- [Background] Vernon WB, Atkins JM, Stewart RD. Hyperphosphatemia from lipid emulsion in a patient on total parenteral nutrition. JPEN J Parenter Enteral Nutr. 1988 Jan-Feb;12(1):84-7. doi: 10.1177/014860718801200184. PMID 3125363
- [Background] Nyirenda MJ, Tang JI, Padfield PL, Seckl JR. Hyperkalaemia. BMJ. 2009 Oct 23;339:b4114. doi: 10.1136/bmj.b4114. No abstract available. PMID 19854840
- [Background] Mendoza J, Legido J, Rubio S, Gisbert JP. Systematic review: the adverse effects of sodium phosphate enema. Aliment Pharmacol Ther. 2007 Jul 1;26(1):9-20. doi: 10.1111/j.1365-2036.2007.03354.x. PMID 17555417
- [Background] Leaf DE, Wolf M. A physiologic-based approach to the evaluation of a patient with hyperphosphatemia. Am J Kidney Dis. 2013 Feb;61(2):330-6. doi: 10.1053/j.ajkd.2012.06.026. Epub 2012 Aug 30. PMID 22938849
- [Background] Eliacik E, Yildirim T, Sahin U, Kizilarslanoglu C, Tapan U, Aybal-Kutlugun A, Hascelik G, Arici M. Potassium abnormalities in current clinical practice: frequency, causes, severity and management. Med Princ Pract. 2015;24(3):271-5. doi: 10.1159/000376580. Epub 2015 Mar 11. PMID 25766276
- [Background] Busch RA, Curtis CS, Leverson GE, Kudsk KA. Use of Piggyback Electrolytes for Patients Receiving Individually Prescribed vs Premixed Parenteral Nutrition. JPEN J Parenter Enteral Nutr. 2015 Jul;39(5):586-90. doi: 10.1177/0148607113518583. Epub 2014 Jan 3. PMID 24390715
- [Background] Kelly DG. Guidelines and available products for parenteral vitamins and trace elements. JPEN J Parenter Enteral Nutr. 2002 Sep-Oct;26(5 Suppl):S34-6. doi: 10.1177/014860710202600510. No abstract available. PMID 12216718